CLINICAL TRIAL: NCT00431730
Title: Is There a Difference in Flicker Induced Vasodilatation Between Smokers and Non-Smokers?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjäeger-Mayrl, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: OPHT-121203
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Ocular Physiology; Retina; Blood Flow Velocity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: flicker light stimulation

SUMMARY:
Habitual smoking is associated with an increased risk of coronary artery disease, cerebral and peripheral vascular disease, including ocular diseases like age-related macular degeneration or diabetic retinopathy. Data of a recent study performed in the investigators lab revealed abnormal choroidal blood flow regulation in chronic smokers as compared to age-matched non-smoking subjects during isometric exercise. However, no information is yet available about the regulation of retinal vascular tone in habitual smokers.

Thus, in the current study, the investigators set out to investigate whether the regulation of retinal vessels diameters is affected in habitual smokers. It has been shown in several reports that stimulation with diffuse luminance flicker, increases retinal arterial and venous diameters, indicating for the ability of the retina to adapt to changing metabolic demands. In the current study we use this effect as a tool to investigate whether the flicker induced vasodilatation is affected in habitual smokers. This would indicate for an impaired vascular regulation process in smokers.

ELIGIBILITY:
Inclusion Criteria:

* 24 subjects aged between 18 and 35 years, nonsmokers (since at least 2 years)
* 24 subjects aged between 18 and 35 years, smokers (at least 10 cigarettes/day since 2 years)
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropy >= 3 dpt

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Flicker response (Retinal vessel analyzer, Laser Doppler Velocimetry)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of CLinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria